CLINICAL TRIAL: NCT03040024
Title: A Randomized Placebo-controlled Pilot Study of Single-dose Intraoperative Ketamine for the Prevention of Delirium in Otolaryngeal Cancer Surgery Patients
Brief Title: Delirium Prevention With Ketamine in Ear, Nose, and Throat (ENT) Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Halted due to COVID 19; we believe we have adequate data for analysis
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Amit Prabhakar, Assistant Professor, Emory University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: IRB00086609
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Results first posted 2021-03-19 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Otolaryngeal Cancer
Keywords: Anesthesiology
MeSH Terms: interventions — Ketamine; Saline Solution; Electroencephalography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketamine 0.5 mg/kg (Experimental): Participants undergoing surgery for otolaryngeal cancer will be randomized to receive one dose of IV ketamine at 0.5 mg/kg.
  Interventions: Drug: Ketamine; Device: Electroencephalogram (EEG)
- Ketamine 1.0 mg/kg (Experimental): Participants undergoing surgery for otolaryngeal cancer will be randomized to receive one dose of IV ketamine at 1.0 mg/kg.
  Interventions: Drug: Ketamine; Device: Electroencephalogram (EEG)
- Placebo (Placebo Comparator): Participants undergoing surgery for otolaryngeal cancer will be randomized to receive one dose of IV saline/placebo.
  Interventions: Drug: Placebo; Device: Electroencephalogram (EEG)

INTERVENTIONS:
Drug: Ketamine — Ketamine will be administered intravenously after administration of general anesthesia and prior to the first surgical incision.
  Arms: Ketamine 0.5 mg/kg; Ketamine 1.0 mg/kg
Drug: Placebo — Placebo will be administered intravenously after administration of general anesthesia and prior to the first surgical incision.
  Other Names: Saline Solution
  Arms: Placebo
Device: Electroencephalogram (EEG) — A processed EEG device will be used during the surgical procedure to gather raw EEG data for off line analysis among patients developing post-operative delirium.

SUMMARY:
The goal of this prospective randomized double blinded placebo controlled study is to investigate if a single dose of ketamine in addition to standard anesthesia will reduce the risk of delirium in otolaryngeal cancer patients postoperatively. Ketamine's effect on post-operative pain and opioid use will be measured as well. Electroencephalogram (EEG) will be utilized during the surgical procedure to evaluate its potential as a possible predictive device for delirium.

DETAILED DESCRIPTION:
This is a single center prospective randomized double blinded placebo controlled study.

The primary aim of the study is to optimize the intraoperative treatment protocol for head and neck cancer patients to reduce the incidence of delirium and associated postoperative cognitive dysfunction. Secondary aims are to determine the dose response relationship for intraoperative ketamine and delirium reduction, determine if a single dose of ketamine will reduce post-operative pain and opioid requirements, determine if raw electroencephalogram (EEG) data can predict postoperative delirium during general anesthesia, and to evaluate length of intensive care unit (ICU) and length of hospital stay.

Participants will be randomized to one of three groups after administration of general anesthesia; one dose of .5 mg/kg intravenous (IV) Ketamine, 1.0 mg/kg of IV Ketamine, or IV placebo.

An EEG will be used during the surgical procedure to gather raw data for off line analysis among patients developing post-operative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of otolaryngeal cancer and undergoing surgery with general anesthesia
* Competent to provide informed consent

Exclusion Criteria:

* Emergency surgery
* Monitored Anesthesia Care (i.e., regional anesthesia alone without plans for general anesthesia)
* Surgery involving the eye, eyebrow, forehead, or frontal scalp near the sensor placement
* Poor health literacy
* Allergy, or have experienced any drug reaction to ketamine
* Pregnant or lactating
* Currently in active alcohol withdrawal
* Taking buprenorphine for chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Moll, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg | Placebo
Started | 21 | 26 | 24
Completed | 21 | 24 | 23
Not Completed | 0 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg | Placebo | Total
Number analyzed (Participants) | 21 | 26 | 24 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.6) | 64.6 (12.4) | 64.5 (11.5) | 64.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 8 | 25
  Male | 12 | 18 | 16 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 20 | 26 | 24 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 4 | 10
  White | 18 | 21 | 20 | 59
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 26 | 24 | 71

OUTCOME MEASURES:

1. Primary Outcome: Change in Confusion Assessment Method fo Intensive Care Unit (CAM-ICU) Delirium Score
Description: The CAM-ICU assesses four features: 1) acute change or fluctuation in mental status from baseline, 2) inattention, 3) altered level of consciousness, and 4) disorganized thinking. The measure reports whether a participant meets criteria for delirium by summing the number of features answered as "present". Feature 1 plus 2 and either 3 or 4 present = delirium positive. Results are expressed as number of participants with or without delirium at each time frame.
Time Frame: Baseline (Up to 30 minutes after PACU arrival), Post Operative (PACU discharge up to 6 hours)
Population: Unable to collect data in 15 participants. N=12: Provider not available. N=2 No PACU. N=1 Physician Decision (withdrawal)
Measure: Count of Participants; unit: Participants
Groups:
- Ketamine 0.5 mg/kg: Participants undergoing surgery for otolaryngeal cancer were randomized to receive one dose of IV ketamine at 0.5 mg/kg.
  Ketamine: Ketamine was administered intravenously after administration of general anesthesia and prior to the first surgical incision.
  Electroencephalogram (EEG): A processed EEG device was used during the surgical procedure to gather raw EEG data for off line analysis among patients developing post-operative delirium.
- Ketamine 1.0 mg/kg: Participants undergoing surgery for otolaryngeal cancer were randomized to receive one dose of IV ketamine at 1.0 mg/kg.
  Ketamine: Ketamine was administered intravenously after administration of general anesthesia and prior to the first surgical incision.
  Electroencephalogram (EEG): A processed EEG device was used during the surgical procedure to gather raw EEG data for off line analysis among patients developing post-operative delirium.
- Placebo: Participants undergoing surgery for otolaryngeal cancer were randomized to receive one dose of IV saline/placebo.
  Placebo: Placebo was administered intravenously after administration of general anesthesia and prior to the first surgical incision.
  Electroencephalogram (EEG): A processed EEG device was used during the surgical procedure to gather raw EEG data for off line analysis among patients developing post-operative delirium.
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg | Placebo
Number analyzed (Participants) | 17 | 22 | 17
Participants
  Delirium CAM-ICU Score at PACU Arrival | 11 | 9 | 9
  No Delirium CAM-ICU Score at PACU Arrival | 6 | 13 | 10
  Delirium CAM-ICU Score at PACU Discharge | 6 | 5 | 2
  No Delirium CAM-ICU Score at PACU Discharge | 11 | 17 | 15

2. Secondary Outcome: Change in Behavioral Pain Scale (Non-Intubated) Score
Description: The Behavioral Pain Scale. Scores range from 3 (no pain) to 12 (maximum pain).
Time Frame: Post Operation (Up to 6 Hours), Post Operation Day 0
Population: Unable to collect information for this outcome. The investigators collected the pain scales from the EMR. The BPS was not routinely collected in the hospital and they only report Visual analog scale (VAS).
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change in Pain Level Assessed by the Visual Analog Scale (VAS) Score
Description: Scores range from 0 (no pain) to 10 (worst pain).
Time Frame: Baseline, Post Surgery (PACU), Post surgery (POD 0), Post surgery (POD 1), Post surgery (POD 2), Post surgery (POD 3), Post surgery (follow up visit - Up to 6 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg | Placebo
Number analyzed (Participants) | 21 | 26 | 24
units on a scale
  Baseline Pain Level assessed by the Visual Analog Scale (VAS) Score | 3.50 (3.25) | 4.36 (2.94) | 2.30 (2.88)
  Pain Level assessed by the Visual Analog Scale (VAS) Score Post surgery (PACU) | 1.00 (2.45) | 2.56 (3.28) | 1.63 (3.11)
  Pain Level assessed by the Visual Analog Scale (VAS) Score Post surgery (POD 0) | 4.76 (3.86) | 4.22 (3.24) | 3.62 (3.74)
  Pain Level assessed by the Visual Analog Scale (VAS) Score Post surgery (POD 1) | 3.93 (2.76) | 3.72 (2.55) | 3.52 (2.42)
  Pain Level assessed by the Visual Analog Scale (VAS) Score Post surgery (POD 2) | 2.47 (2.52) | 2.81 (2.51) | 3.38 (2.62)
  Pain Level assessed by the Visual Analog Scale (VAS) Score Post surgery (POD 3) | 3.08 (2.94) | 3.35 (2.15) | 3.41 (2.20)
  Pain Level assessed by the Visual Analog Scale Score Post surgery (follow up visit - Up to 6 weeks) | 2.3 (2.58) | 3.09 (2.68) | 3.00 (2.60)

4. Secondary Outcome: Change in Mini Cog Score
Description: The Mini-Cog is a 3-minute instrument that can increase detection of cognitive impairment. A score ranging from 0-2 indicates positive screen for dementia. A score ranging from 3-5 indicates negative screen for dementia.
Time Frame: Baseline, Post Surgery (Up to 6 Weeks)
Population: The number of participants is different from participant flow because some of the subjects did not complete the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg | Placebo
Number analyzed (Participants) | 20 | 25 | 24
Participants
  Baseline Mini Cog Score- Positive Screen | 2 | 5 | 6
  Baseline Mini Cog Score- Negative Screen | 18 | 20 | 18
  Mini Cog Score Post surgery (Up to 6 weeks) - Positive Screen: number analyzed (Participants) | 20 | 23 | 20
  Mini Cog Score Post surgery (Up to 6 weeks) - Positive Screen | 3 | 0 | 3
  Mini Cog Score Post surgery (Up to 6 weeks) - Negative Screen: number analyzed (Participants) | 20 | 23 | 20
  Mini Cog Score Post surgery (Up to 6 weeks) - Negative Screen | 17 | 23 | 17

5. Secondary Outcome: Change in Mini-Mental Status Examination (MMSE) Score
Description: The MMSE is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. Any score greater than or equal to 24 points (out of 30) indicates a normal cognition. Below this (0-24), scores can indicate cognitive impairment.
Time Frame: Baseline, Post Surgery (Up to 6 Weeks)
Population: This assessment was not completed for some subjects, and that is the reason why the number analyzed is different from the overall number analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg | Placebo
Number analyzed (Participants) | 20 | 25 | 24
Participants
  Normal Baseline MMSE Score (25-30) | 18 | 22 | 22
  Cognitive Impairment Baseline MMSE Score (0-24) | 2 | 3 | 2
  Normal Post surgery (Up to 6 weeks) MMSE Score (25-30): number analyzed (Participants) | 20 | 23 | 20
  Normal Post surgery (Up to 6 weeks) MMSE Score (25-30) | 17 | 23 | 16
  Cognitive Impairment Post surgery (Up to 6 weeks) MMSE Score (0-24): number analyzed (Participants) | 20 | 23 | 20
  Cognitive Impairment Post surgery (Up to 6 weeks) MMSE Score (0-24) | 3 | 0 | 4

6. Secondary Outcome: Change in Cognitive Failure Questionnaire (CFQ) Score
Description: The CFQ is a 25-item self-report measure of failures in attention, perception, memory, and action. Participants are asked to indicate on a 5-point scale how often they have experienced each failure in the past months, from 0 (never) to 5 (very often). Scores range from 0 to 100 a higher score indicating more failures in attention.
Time Frame: Baseline, Post Surgery (Up to 6 Weeks)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg | Placebo
Number analyzed (Participants) | 20 | 25 | 24
score on a scale
  Baseline CFQ Score: number analyzed (Participants) | 18 | 25 | 24
  Baseline CFQ Score | 27 [21 to 38] | 34 [22 to 40] | 30 [21.5 to 38.5]
  CFQ Score Post surgery (Up to 6 weeks): number analyzed (Participants) | 20 | 23 | 20
  CFQ Score Post surgery (Up to 6 weeks) | 29 [23 to 35] | 30 [15 to 40] | 29 [23 to 37]

7. Secondary Outcome: Post Operative Narcotics Use
Description: The total amount of narcotics used measured in morphine milligram equivalents (MME).
Time Frame: Post Intervention (Intraoperative), Post Intervention (POD 0), Post Intervention (POD 1),Post Intervention (POD 2),Post Intervention (POD 3), Post Intervention (Follow up visit-up to 6 weeks post intervention)
Population: The population is different at 6 weeks post intervention because this outcome was not completed for some participants at that time point.
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents (MME)
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg | Placebo
Number analyzed (Participants) | 21 | 26 | 24
morphine milligram equivalents (MME)
  Post Intervention (Intraoperative) | 13.3 [6.7 to 13.33] | 13.3 [10.0 to 20.0] | 13.33 [8.75 to 16.00]
  Post Intervention (POD 0) | 7.1 [0 to 11.9] | 6.67 [0 to 11.9] | 6.18 [3.3 to 15.1]
  Post Intervention (POD 1) | 35 [10.7 to 57.7] | 41.5 [27.1 to 91.4] | 42.9 [25.7 to 51.4]
  Post Intervention (POD 2) | 8.59 [2.0 to 53.8] | 25.7 [10.0 to 78.6] | 41.9 [17.3 to 51.4]
  Post Intervention (POD 3) | 19.8 [0.0 to 40.8] | 34.3 [2.0 to 50.7] | 34.3 [17.1 to 44.9]
  Post Intervention (Follow up visit-up to 6 weeks): number analyzed (Participants) | 21 | 23 | 21
  Post Intervention (Follow up visit-up to 6 weeks) | 0 [0 to 8.6] | 0 [0 to 38.4] | 0 [0 to 25.7]

8. Secondary Outcome: Associations of Intraoperative EEG Patterns With PACU Delirium
Description: The investigators compared the relative beta power derived from the normalized power spectral density (PSD) in patients with and without PACU delirium (positive and negative delirium). Only a total of 38 EEGs with sufficient quality were analyzed. Results are expressed in percentage of cumulative power. A higher beta power correlates with worse outcome. Averages and standard deviations are shown.
Time Frame: Intraoperative EEG and delirium during PACU stay
Population: Only a total of 38 EEGs with sufficient quality were analyzed
Measure: Mean (Standard Deviation); unit: Percentage of cumulative power
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg | Placebo
Number analyzed (Participants) | 18 | 9 | 11
Percentage of cumulative power
  Positive Delirium for PACU: number analyzed (Participants) | 6 | 5 | 2
  Positive Delirium for PACU | 10.0 (5.0) | 7.0 (5.0) | 7.0 (6.0)
  Negative Delirium for PACU: number analyzed (Participants) | 12 | 4 | 9
  Negative Delirium for PACU | 7.0 (1.0) | 5.0 (6.0) | 6.0 (4.0)

ADVERSE EVENTS:
Time Frame: The research team monitored subjects randomized and treated in the study for adverse events related to the research through the final study visit in the ENT clinic that occurred from 2 to 6 weeks post-operatively.
Description: If the change from baseline was considered by the investigator to be part of the normal fluctuations of an underlying disease process, this was not reported as an adverse event (AE). If the change in baseline was considered by the investigator to be an untoward medical occurrence different from the standard of care, this medical occurrence was reported as an AE.
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 1/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 4/21 | 9/26 | 2/24
Other Adverse Events (participants affected / at risk) | 3/21 | 5/26 | 4/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine 0.5 mg/kg (N=21) | Ketamine 1.0 mg/kg (N=26) | Placebo (N=24)
Delirium (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial artery clot (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Surgical wound dehiscence (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid injury (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Post-operative wound abscess (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bilateral MCA; PCA transcortical acute infarcts (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
NSTEMI (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
Partial flap necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Exposed tendon of left forearm free flap (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine 0.5 mg/kg (N=21) | Ketamine 1.0 mg/kg (N=26) | Placebo (N=24)
Agitation (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Transient left sided weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (General disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Restlessness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT03040024/Prot_SAP_000.pdf